CLINICAL TRIAL: NCT01224886
Title: In French AGIR Means to Get Into Action. This is the Generic Title of Our Study.
Brief Title: Age and Insulin Resistance
Acronym: AGIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Francesca Amati, Associate Professor, University of Lausanne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGIR; Protocol 188/10 (Other: Ethics committee)
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Physical Inactivity; Aging
Keywords: Aging; Insulin resistance; Ectopic lipids; Obesity; Exercise; Physical activity; Oxidative capacity; Diabetes; Metabolic syndrome
MeSH Terms: conditions — Obesity; Sedentary Behavior; Insulin Resistance; Motor Activity; Diabetes Mellitus; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sedentary obese (Experimental)
  Interventions: Behavioral: Physical activity
- Sedentary normal weight (Experimental)
  Interventions: Behavioral: Physical activity
- Athletes (No Intervention)

INTERVENTIONS:
Behavioral: Physical activity — Supervised exercise intervention
  Arms: Sedentary normal weight; Sedentary obese

SUMMARY:
Insulin resistance is a crucial factor for the development of type 2 diabetes and a major health problem for older adults. It is the principal mechanism by which obesity is considered to increase the risk for type 2 diabetes and is a key feature of the metabolic syndrome. The elevated prevalence of obesity and type 2 diabetes in the older population has important consequences on the morbidity and mortality as well as on the economic burden on society. Controversy currently exists as to whether or not aging contributes to insulin resistance. Many potential factors confound the association between aging and insulin resistance, including obesity and physical inactivity.

Ectopic lipid depositions, defined as an excess accumulation of triglycerides in non adipose tissues such as in the liver (intrahepatic lipids) and within the muscle fibers (intramyocellular lipids), are positively associated with obesity and insulin resistance. Furthermore, the accumulation of intracellular lipids is often cited as being a key determinant in the underlying mechanisms of insulin resistance. In addition of playing an important role in obesity and type 2 diabetes, these ectopic fat depositions are also observed in common conditions such as aging and physical inactivity.

The intervention trial will test in skeletal muscle, liver and heart of sedentary obese volunteers, normal weight volunteers and masters athletes, the overall hypotheses that exercise improvement of fat oxidation capacity and/or decrease of damaging fat metabolites is a primary factor that predicts the improvement in insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80
* Sedentary or highly trained
* BMI 18-40
* Non-Smoker
* Normal glucose tolerance or impaired glucose tolerance
* Willingness to comply with the protocol

Exclusion Criteria:

* Contraindication to moderate exercise or clinical conditions precluding from joining an exercise program, such as clinically significant cardiovascular disease, peripheral vascular disease, uncontrolled hypertension, neurological or orthopedic disease
* Recent weight loss or weight gain
* Known diabetes
* Known drugs to affect glucose homeostasis such as nicotinic acid, glucocorticoids
* Severe anemia or lipid disturbances, hepatic or renal disease
* Recent history of cancer
* Hypothyroidism
* Recent hormone replacement therapy
* Known allergy to lidocaine or other local anesthetic
* Positive stress test
* Active alcohol or substance abuse

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 0-4 months
Ectopic lipids | 0-4 months
Oxidative capacity | 0-4 months

SECONDARY OUTCOMES:
Body composition | 0-4 months
Metabolic flexibility | 0-4 months
Exercise efficiency | 0-4 months
Physical fitness | 0-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Amati, MD,PhD, Principal Investigator — University of Lausanne
Locations (2):
- Switzerland (2):
  - University of Bern, Bern
  - UNIL and CHUV, Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greggio C, Jha P, Kulkarni SS, Lagarrigue S, Broskey NT, Boutant M, Wang X, Conde Alonso S, Ofori E, Auwerx J, Canto C, Amati F. Enhanced Respiratory Chain Supercomplex Formation in Response to Exercise in Human Skeletal Muscle. Cell Metab. 2017 Feb 7;25(2):301-311. doi: 10.1016/j.cmet.2016.11.004. Epub 2016 Dec 1. PMID 27916530
- [Result] Broskey NT, Boss A, Fares EJ, Greggio C, Gremion G, Schluter L, Hans D, Kreis R, Boesch C, Amati F. Exercise efficiency relates with mitochondrial content and function in older adults. Physiol Rep. 2015 Jun;3(6):e12418. doi: 10.14814/phy2.12418. PMID 26059033
- [Result] Broskey NT, Greggio C, Boss A, Boutant M, Dwyer A, Schlueter L, Hans D, Gremion G, Kreis R, Boesch C, Canto C, Amati F. Skeletal muscle mitochondria in the elderly: effects of physical fitness and exercise training. J Clin Endocrinol Metab. 2014 May;99(5):1852-61. doi: 10.1210/jc.2013-3983. Epub 2014 Jan 17. PMID 24438376
- [Result] Broskey NT, Daraspe J, Humbel BM, Amati F. Skeletal muscle mitochondrial and lipid droplet content assessed with standardized grid sizes for stereology. J Appl Physiol (1985). 2013 Sep 1;115(5):765-70. doi: 10.1152/japplphysiol.00063.2013. Epub 2013 Jun 20. PMID 23788579
- [Result] Amati F, Broskey NT, Carnero EA. Evidence of systematic and proportional error in a widely used glucose oxidase analyser: impact for clinical research? Clin Endocrinol (Oxf). 2014 May;80(5):768-70. doi: 10.1111/cen.12274. Epub 2013 Jul 19. No abstract available. PMID 23800101